CLINICAL TRIAL: NCT05458986
Title: A Pilot Video Intervention to Decrease Fear of Colonoscopy in a Safety-Net Healthcare System
Brief Title: A Video Intervention to Decrease Patient Fear of Colonoscopy After a Positive Fecal Immunochemical Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RG1122309; NCI-2022-05223 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10950 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2022-07-01; First posted 2022-07-14 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Practice Guidelines as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (educational video) (Experimental): Patients watch an educational video about the importance of abnormal FIT results, the implications if follow-up colonoscopy is not completed, and demonstrate the steps to complete a colonoscopy.
  Interventions: Other: Media Intervention; Other: Questionnaire Administration
- Arm 2 (usual care) (Active Comparator): Patients receive usual care and do not watch the educational video.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Media Intervention — Watch an educational video
  Arms: Arm 1 (educational video)
Other: Best Practice — Receive usual care
  Arms: Arm 2 (usual care)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial compares an educational video intervention versus usual care of no video intervention in decreasing patient fear of a colonoscopy procedure after receiving a positive fecal immunochemical test (FIT). The lack of a follow-up colonoscopy after an abnormal FIT result is associated with an increased risk of colorectal cancer mortality, advanced-stage colorectal cancer, among other complications, compared to the completion of a follow-up colonoscopy. An educational video may reduce patient fear and increase knowledge, self-efficacy, and intent to complete a colonoscopy compared to the usual care of no video intervention.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients watch an educational video about the importance of abnormal FIT results, the implications if follow-up colonoscopy is not completed, and demonstrate the steps to complete a colonoscopy.

ARM 2: Patients receive usual care and do not watch the educational video.

After completion of study, patients are followed for 12 months after their abnormal FIT result.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75
* Have an assigned primary care provider in our partnering safety-net health system
* Have a billable primary care encounter between 2019-2022
* Have an abnormal FIT result for colorectal cancer (CRC) screening without a colonoscopy within 1 year
* Ability to communicate in English due to initial videos being available in English

Exclusion Criteria:

* Adults < age 45 or > age 75
* Patients who receive care at other University of Washington (UW) medicine sites (non-safety-net patients)
* Individuals without a primary care encounter between 2019-2022
* Individuals whose primary language is not English

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by study accrual | Up to 12 months post-abnormal fecal immunochemical test (FIT) result
  Feasibility will be measured by recruitment as the proportion of invited participants who consent and complete the pilot study.
Feasibility: number of contacts needed to reach target enrollment | Up to 12 months post-abnormal FIT result
  Feasibility will be measured by recruitment as the number of contacts required to reach target enrollment.
Feasibility: time to reach recruitment | Up to 12 months post-abnormal FIT result
  Feasibility will be measured by recruitment as the time required to reach target enrollment. Time to reach recruitment target will be measured in days and described using medians and interquartile range (IQR).
Acceptability of the video intervention assessed by a survey | Up to 12 months post-abnormal FIT result
  Intervention arm patients will complete a post-intervention survey to assess acceptability of the intervention using the Acceptability of Intervention Measure (AIM), a 4-item measure. Items are rated on a 5-point Likert Scale (1, completely disagree; 5, completely agree). Mean scores will be calculated to generate an average AIM score, where higher scores will indicate higher levels of acceptability.
Incidence of fear related to colonoscopy | Up to 12 months post-abnormal FIT result
  Intervention arm patients will complete a pre- and post-intervention survey that will include questions about fear of colonoscopy. Usual care patients will complete a baseline survey on the same measures. Fear will be assessed using Manne's 6-item fear of colonoscopy scale. Items are rated on a 5-point Likert scale (1, not at all fearful; 5, extremely fearful). Mean scores will be calculated to generate average fear per participant, with higher scores indicating higher levels of fear.
Knowledge about colonoscopy | Up to 12 months post-abnormal FIT result
  Intervention arm patients will complete a pre- and post-intervention survey that will include questions about knowledge about colon cancer screening. Usual care patients will complete a baseline survey on the same measures. Knowledge will be measured using 8 validated questions. Incorrect answers will be scored as 0 and correct answers scored as 1. Higher scores will indicate higher levels of knowledge.
Self-efficacy related to colonoscopy | Up to 12 months post-abnormal FIT result
  Intervention arm patients will complete a pre- and post-intervention survey that will include questions about self-efficacy related to a colonoscopy. Usual care patients will complete a baseline survey on the same measures. Self-efficacy will be assessed by adopting an 8-item self-efficacy scale for colonoscopy completion in patients with inflammatory bowel diseases and responses will be recorded on a 5-point scale. Higher scores will indicate higher levels of self-efficacy.
Intent to complete a colonoscopy | Up to 12 months post-abnormal FIT result
  Intervention arm patients will complete a pre- and post-intervention survey that will include questions about intent to complete a colonoscopy. Usual care patients will complete a baseline survey on the same measures. Intent will be measured using a single validated question on a nominal scale with 5 options. Responses will be dichotomized to affirmative intent (definitely will do, will do) or uncertain intent (don't know, will not do, and definitely will not do).

SECONDARY OUTCOMES:
Incidence of completed colonoscopies | At 6 months post randomization
  Through review of the electronic health records (EHR), the investigators will determine rates of completed colonoscopy 6 months after randomization to assess preliminary efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Issaka, MD, MAS, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT05458986/ICF_000.pdf